CLINICAL TRIAL: NCT05745571
Title: Molecular Pathways of Cardiac Remodellation in Patients With Acute and Chronic Left Ventricular Disfunction (HFrEF)
Brief Title: Molecular Pathways of Cardiac Remodellation in Patients With Acute and Chronic Left Ventricular Disfunction
Acronym: HFrEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Liuzzo Giovanna, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2291
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure; Ischemic Cardiomyopathy
Keywords: Ejection Fraction (EF); Sympathetic nervous system (SNS); Renin-angiotensin-aldosterone system (RAAS)
MeSH Terms: conditions — Heart Failure | interventions — Blood Specimen Collection; Proteins

STUDY DESIGN:
Intervention Model Description: Our study will be interventional, prospective, and single-center. At the time of enrollment in the study, peripheral blood will be drawn, then patients will be recalled for follow-up visits at 1 and 6 months, during which new venous blood draws will be performed, together with the echocardiographic examination. Patients will undergo the treatment required by the current and most recent guidelines for heart failure and adherence to this study will not involve any modification of the current therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with acute coronary syndrome (Other): 30 patients admitted to our hospital with the diagnosis of STEMI-type ACS and ejection fraction ≤ 35% on echocardiographic evaluation
  Interventions: Other: Blood sample
- Patients with non-ischaemic dilated cardiomyopathy (Other): 30 patients with non-ischaemic dilated cardiomyopathy and ejection fraction ≤35% on echocardiographic evaluation
  Interventions: Other: Blood sample
- Patients diagnosed with STEMI-type ACS (Other): Patients diagnosed with STEMI-type ACS and ejection fraction > 50% on echocardiographic evaluation
  Interventions: Other: Blood sample
- Controls (Other): Controls with normal left ventricular contractile function
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — The study foresees a phase of patient recruitment, in which, in the hours immediately following the blood sampling, the isolation of the PBMCs, their incubation and cytofluorimetric analysis will be carried out and the conservation of the material to be analyzed subsequently by molecular biology and immunochemistry.
  Other Names: Molecular pathway and protein

SUMMARY:
Chronic heart failure represents an extremely complex clinical syndrome, defined as the inability of the heart muscle to generate a volume adequate to the metabolic needs of peripheral tissues, or to do so only in the face of high filling pressures intracavity. Heart failure is one of the leading causes of mortality and morbidity in Western countries.

Despite advances in the therapeutic field, the prognosis of patients with heart failure of ischemic and non-ischaemic aetiology still remains unfavorable, with a mortality rate of 50% 5 years after the first hospitalization.Therefore, a deeper understanding of the pathophysiological mechanisms involved in heart failure and adverse ventricular remodeling is essential.

DETAILED DESCRIPTION:
The study will be interventional, prospective, and single-center. Partecipants will be divided into three groups:

1. 30 partecipants admitted to our hospital with the diagnosis of STEMI-type ACS and ejection fraction ≤ 35% on echocardiographic evaluation
2. 30 partecipants with non-ischaemic dilated cardiomyopathy and ejection fraction ≤35% on echocardiographic evaluation
3. 15 partecipants diagnosed with STEMI-type ACS and ejection fraction > 50% on echocardiographic evaluation
4. 15 controls with normal left ventricular contractile function. The study foresees a phase of patient recruitment, in which, in the hours immediately following the blood sampling, the isolation of the PBMCs, their incubation and cytofluorimetric analysis will be carried out and the conservation of the material to be analyzed subsequently by molecular biology and immunochemistry.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the Gemelli Polyclinic with acute coronary syndromes and heart disease;
* patients admitted to our polyclinic with the diagnosis of SCA type STEMI and ejection fraction ≤ 35% at echocardiographic evaluation;
* patients with non-ischemic dilated cardiomyopathy and ejection fraction ≤ 35% at echocardiographic evaluation;
* patients diagnosed with SCA type STEMI and ejection fraction > 50% at echocardiographic evaluation;

Exclusion Criteria:

* evidence of inflammatory or infectious disease;
* malignancy, or immunological or hematologic disorders;
* treatment with anti-inflammatory drugs other than low-dose aspirin;
* age > 85 years;
* recent surgery (within one month);
* advanced chronic kidney disease (eGFR MDRD-4 <30 ml/min./1.73m2).

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Study of molecular pathways involved in acute cardiac dysfunction and cardiac remodelling | 10 months
  Gene expression assessment of molecular pathways involved in acute cardiac dysfunction and cardiac remodelling underlying reduced ejection fraction heart failure (HFrEF).
  Evaluation of protein expression of specific markers by means of cytofluorimetric and immunochemical methods, the choice of which will be made after the analysis of the molecular gene patterns most commonly represented in patients with left ventricular contractile dysfunction.The study includes a patient recruitment phase, in which the isolation of PBMCs, their incubation and cytofluorimetric analysis will be carried out in the hours immediately following the blood sampling, and the material will be stored for subsequent analysis by molecular biology and immunochemistry analysis.

SECONDARY OUTCOMES:
Experiments to identify possible molecular targets for future studies | 6 months
  Carrying out mechanistic experiments to verify the biological significance of altering specific molecular patterns and identifying possible molecular targets for subsequent studies.
  For these future studies, it is planned to store material for retrospective analysis by molecular biology and immunochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No